CLINICAL TRIAL: NCT06838273
Title: A Phase III Randomized Study of BL-B01D1 in Combination With Osimertinib Versus Osimertinib as First-Line Treatment in Patients With EGFR-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of BL-B01D1 in Combination With Osimertinib Versus Osimertinib as First-Line Treatment in Patients With EGFR-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-308
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 in Combination with Osimertinib (Experimental): Participants receive BL-B01D1 in Combination with Osimertinib for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: Osimertinib
- Osimertinib (Active Comparator): Participants receive Osimertinib for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1 in Combination with Osimertinib
Drug: Osimertinib — Oral administration, 80mg daily for a cycle of 3 weeks.
  Arms: BL-B01D1 in Combination with Osimertinib
Drug: Osimertinib — Oral administration, 80mg daily for a cycle of 3 weeks.
  Arms: Osimertinib

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in combination with osimertinib versus osimertinib as first-Line treatment in patients with EGFR-mutated locally advanced or metastatic Non-small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Age ≥18 years old;
3. Expected survival time ≥3 months;
4. Patients with unresectable or radical radiotherapy for locally advanced non-small cell lung cancer;
5. Documentation of EGFR sensitive mutations detected from tumor tissue or blood samples;
6. Consent to provide archived tumor tissue samples or fresh tissue samples of primary or metastatic lesions at or after diagnosis for testing, including EGFR mutation type;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. The organ function level must meet the requirements on the premise that blood transfusion and colony-stimulating factor are not allowed within 14 days before the screening period;
12. Urinary protein ≤2+ or < 1000mg/24h;
13. For premenopausal women of childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and the patient must not be lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Previous histologic or cytological evidence of small cell or mixed small/non-small cell components;
2. Patients with previous systemic therapy;
3. Patients had received EGFR-TKI therapy;
4. Studies received radical radiotherapy, major surgery, and large area radiotherapy within 4 weeks before randomization;
5. History of severe heart disease and cerebrovascular disease;
6. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
7. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
8. Were diagnosed with active malignancy within 3 years before randomization;
9. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
10. Patients with poor glycemic control;
11. A history of ILD requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis, or a suspicion of such disease;
12. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
13. Patients with active central nervous system metastasis;
14. Had a severe infection within 4 weeks before randomization;
15. Patients with massive or symptomatic effusions or poorly controlled effusions;
16. Imaging examination showed that the tumor had invaded or enveloped the large blood vessels in the abdomen, chest, neck, and pharynx;
17. Serious unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
18. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
19. Patients with a history of inflammatory bowel disease, extensive bowel resection, immune enteritis, intestinal obstruction or chronic diarrhea;
20. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of BL-B01D1;
21. Had autologous or allogeneic stem cell transplantation history;
22. Human immunodeficiency virus antibody positive, active hepatitis B virus infection or hepatitis C virus infection;
23. A history of severe neurological or psychiatric illness;
24. Received other unmarketed investigational drugs or treatments within 4 weeks before randomization;
25. Subjects scheduled for vaccination or who received live vaccine within 28 days before study randomization;
26. Other circumstances in which the investigator considered it inappropriate to participate in the trial because of complications or other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 36 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 36 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Objective Response Rate (ORR) | Up to approximately 36 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 36 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 36 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 36 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 36 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China